CLINICAL TRIAL: NCT02156037
Title: Case Management for Underserved Hispanic Type 2 Diabetes Populations
Brief Title: An RCT Evaluation of a Diabetes Dashboard Team Model in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: diabetesdashboardrct
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes
Keywords: Hispanic; clinical decision support; diabetes; Hba1c; psychosocial
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dashboard team care intervention (Experimental): Dashboard team
  Interventions: Behavioral: Diabetes Dashboard Intervention
- usual diabetes team control (Active Comparator): usual clinical diabetes team with no access to the diabetes dashboard
  Interventions: Behavioral: Usual Diabetes Care

INTERVENTIONS:
Behavioral: Diabetes Dashboard Intervention — The Diabetes Dashboard Intervention Condition involved a program of five, in-person, one-on-one diabetes education and behavior change visits with a diabetes nurse or diabetes dietician, scheduled at baseline, two weeks, one month, three months, and six months post-enrollment.
  Arms: dashboard team care intervention
Behavioral: Usual Diabetes Care — The UDC condition was delivered by four bicultural, bilingual diabetes nurses and diabetes dietitians who comprised the clinical site's long-standing, in-house diabetes program.
  Arms: usual diabetes team control

SUMMARY:
To compare a comprehensive diabetes team care condition (IC) involving the diabetes team's use of a "diabetes dashboard" with a usual diabetes team care condition (UDC) that does not have access to the diabetes dashboard.

DETAILED DESCRIPTION:
To compare a usual diabetes care condition (UDC) to a comprehensive diabetes care intervention condition (IC) involving a "diabetes dashboard" clinical decision support tool used by the diabetes team in primary care. The investigators used a parallel-groups randomized design. The diabetes team (i.e., diabetes nurses, diabetes dietitians, and providers) delivered a 5-visit, 6-month intervention to n=199 poorly-controlled (HbA1c >7.5%) Latino T2D patients (mean age=55 years, 60% female) seen at 2 urban community health centers. This intervention was compared to an established, in-house diabetes team care program (n=200) for its impact on blood glucose control and key psychosocial outcomes (diabetes distress, depression, social distress).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older,
* self-identified Hispanic ethnicity,
* diagnosis of T2D,
* HbA1c >7.5%, and
* provider approval given for patient participation

Exclusion Criteria:

* inability to consent,
* pregnant or planning to become pregnant in the next year,
* taking glucocorticoid therapy, or
* having serious psychiatric or medical complications (e.g., late stage diabetes complications, seizures, dementia, psychiatric hospitalization) that would prevent participation in study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Change in HbA1c over 6 months

SECONDARY OUTCOMES:
Diabetes distress | 6 months
  Patient reported diabetes distress associated with Type 2 diabetes and its treatment measured using the PAID scale
Depression | 6 months
  Patient-reported depression status based on the PHQ scale

CONTACTS AND LOCATIONS:
Overall Officials: Garry Welch, PhD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Welch G, Zagarins SE, Santiago-Kelly P, Rodriguez Z, Bursell SE, Rosal MC, Gabbay RA. An internet-based diabetes management platform improves team care and outcomes in an urban Latino population. Diabetes Care. 2015 Apr;38(4):561-7. doi: 10.2337/dc14-1412. Epub 2015 Jan 29. PMID 25633661